CLINICAL TRIAL: NCT04319185
Title: Assisted Peritoneal Dialysis: A Feasibility Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Satellite Healthcare (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SIH123_Assisted PD
Record Dates: First submitted 2020-02-05; First posted 2020-03-24 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: End Stage Kidney Disease; End Stage Renal Disease
Keywords: Peritoneal Dialysis; End Stage Renal Disease (ESRD); End Stage Kidney Disease (ESKD)
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: A mixed-methods feasibility design using quantitative and qualitative techniques will be used to meet the aims of this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): All patients who qualify for the study will receive the intervention
  Interventions: Other: Assistance to perform Peritoneal Dialysis (PD) at home

INTERVENTIONS:
Other: Assistance to perform Peritoneal Dialysis (PD) at home — The patient receives assistance of up to one visit per day for three months depending on the patient's needs, as assessed by the interdisciplinary team, the nephrologist, and the primary investigator or delegate.

SUMMARY:
Patients with End-Stage Kidney Disease (ESKD) wishing to choose Peritoneal Dialysis (PD) may not be able to perform this modality due to advanced age, physical function/dexterity, vision, cognition, mobility, or psychosocial issues. This intervention will seek to test the feasibility of a clinical support model to address these barriers.

Patients identified by their nephrologist as wishing to choose Peritoneal Dialysis (PD), but needing assistance, are referred to the research staff for discussion and consent.

Based on the assessment of the subject's nephrologist, PD staff, and researchers, the subject will receive assistance beyond the standard PD care offered in US dialysis centers. Such assistance will be provided for up to one visit/day, seven days/week, for up to three months. At the end of that time period, the subject will be able to perform PD independently, have identified a care provider, or have planned with his/her nephrologist for an alternative dialysis modality.

DETAILED DESCRIPTION:
A patient identified by his/her nephrologist or the WellBound dialysis staff as a candidate for Peritoneal Dialysis (PD) who meets the inclusion criteria will be referred to the research staff for a discussion of the study and consent. A referral to this program can come from any physician referring to participating centers.

* Each subject consented into the study receives the standard of care education and training for home PD, in addition to the usual insertion of a PD catheter.
* The subject is then transferred to home PD with an individualized assistance plan and research follow-up.
* The subject receives the assistance of up to one visit per day depending on the subject's needs, as assessed by the interdisciplinary team, the nephrologist, and the primary investigator or delegate.
* The assistance will be provided by a research associate who has undergone full training in the PD techniques required to assist the PD subject at home.
* Every 4 weeks the PI or delegate reviews the subject's progress with the nephrologist and nephrology nurse to assess further assistance needs.
* Total assistance of up to 3 months is provided after which the subject is either independent, has a care provider, or has developed a plan with his/her nephrologist for future dialysis care.

ELIGIBILITY:
Inclusion Criteria:

Peritoneal Dialysis (PD) patients identified as needing staff-assistance:

1. Incident peritoneal dialysis patients from participating centers identified by referring nephrologists or PD staff to need the service.

   OR
2. Prevalent PD patients who experience a change in status, making them in need of the service.

Criteria for needing assistance: The patient has one of the following criteria that prevents him or her from an independent PD program as assessed by their nephrologist, and nephrology nurse: advanced age, physical function/dexterity, vision, cognition, mobility, psychosocial issues or other.

Exclusion Criteria:

1. Age less than 18 years
2. Unable to understand English (because of the need to complete the consent form and survey instruments which are available only in English).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-09-11 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
To explore the feasibility of an assisted PD program by assessing the need. | Throughout the study, an average of two years
  Number and proportion of patients needing the service (out of total new starts of PD).
To explore the feasibility of an assisted PD program by assessing the types of need. | Throughout the study, an average of two years
  Categorize types of assisted tasks and length of assistance needed by participants in the program.
To explore the feasibility of an assisted PD program by assessing acceptance. | Throughout the study, an average of two years
  Measure the number and rate of patients recruited.
To explore the feasibility of an assisted PD program by measuring adherence. | Throughout the study, an average of two years
  Measure the number and rate of participants' adherence to and completion of the program.
To explore the feasibility of an assisted PD program by assessing the outcome of participant Peritoneal Dialysis independence. | Throughout the study, average of two years
  Measure the number of patients able to independently continue Peritoneal Dialysis out of all patients referred to the program.
To explore the feasibility of an assisted PD program by assessing any and all adverse events. | Throughout the study, average of two years
  Collect all adverse events during the study.
To explore the feasibility of an assisted PD program by measuring the effect on the program on the participant's ability to maintain PD as the treatment modality. | At 1, 2, 3, 6, and 12 months
  Change in the number of patients who remain on Peritoneal dialysis after assistance as reflected in the dialysis unit records from 1 month to 12 months.
To provide data to estimate the personnel costs of a US assisted PD program. | Aggregated from the start to end of the study (estimated as two years)
  Measurement of the time and, thus, costs of personnel to conduct the assisted PD program.
To provide data to estimate the resources costs of a US assisted PD program. | Aggregated from the start to end of the study (estimated as two years)
  Measurement of all non-personal costs to complete the study.
To identify the demographics of the population in need of assisted PD support. | On referral into the study.
  Assessment of the baseline demographics of the patient as routinely collected in the dialysis record.
To identify the medical history of the population in need of assisted PD support. | Day one on the study
  Assessment of the medical history of the patient as routinely collected in the dialysis record.
To identify the frailty level of the population in need of assisted PD support. | Change from day 1 of home dialysis to 3 months (end of the intervention) .
  Measured by the clinical frailty scale. This ranges from 1 (very fit) to 9 (terminally ill).
To identify the patient activation level of the population in need of assisted PD support. | Change from month 1 through month 3 (end of the intervention).
  Measured by the Patient Activation Measure: PAM-13 survey. This is a 100 point scale with lower scores designating an individual with less ability to manage his/her health and healthcare.
To identify the patient symptom level of the population in need of assisted PD support. | Change from week 1 to month 3 (end of study).
  Measured by the Renal Patient Outcome Scale: IPOS-Renal survey which is composed of 11 questions on renal symptoms and patient issues with higher scores indicating greater distress.
To identify the patient satisfaction with an assisted PD program. | Change from 1 month to the end of the patient's participation in the study (up to 1 year).
  Measured by a simple LIkert Patient Satisfaction Scale ranging from 1 - 5 with higher results indicating greater satisfaction.
To identify the staff's satisfaction with an assisted PD program. | One time at the end of the program (approximately two years).
  Assessed by open ended questions at a staff focus group.

CONTACTS AND LOCATIONS:
Overall Officials: Wael F Hussein, MBBS, Principal Investigator — Satellite Healthcare, Inc.
Locations (6):
- United States (6):
  - Satellite WellBound Emeryville, Emeryville, California
  - Satellite WellBound Fremont, Fremont, California
  - Satellite WellBound Milpitas, Milpitas, California
  - Satellite WellBound Mountain View, Mountain View, California
  - Satellite WellBound San Jose, San Jose, California
  - Satellite WellBound San Mateo, San Mateo, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hussein WF, Chen S, Bennett PN, Atwal J, Abra G, Weinhandl E, Zheng S, Pravoverov L, Schiller B. Description and outcomes of a staff-assisted peritoneal dialysis program in the United States. Perit Dial Int. 2025 Nov;45(6):344-352. doi: 10.1177/08968608241259607. Epub 2024 Jun 17. PMID 38881397
- [Derived] Hussein WF, Bennett PN, Anwaar A, Atwal J, Legg V, Abra G, Zheng S, Pravoverov L, Schiller B. Implementation of a Staff-Assisted Peritoneal Dialysis Program in the United States: A Feasibility Study. Clin J Am Soc Nephrol. 2022 May;17(5):703-705. doi: 10.2215/CJN.00940122. Epub 2022 Apr 5. No abstract available. PMID 35383044